CLINICAL TRIAL: NCT01633086
Title: A Study on the Safety and Efficacy of Nitric Oxide Gel in Subjects With Painful Diabetic Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DMR99-IRB-273
Record Dates: First submitted 2012-05-30; First posted 2012-07-04 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2015-03

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- nitric oxide gel (Active Comparator): 1. st gel: sodium nitrites
  2. nd gel: maleic/ascorbic acids
  Interventions: Drug: nitric oxide gel
- Placebo gel (Placebo Comparator): 1. st gel: phosphate-buffered saline
  2. nd gel: maleic/ascorbic acids
  Interventions: Drug: placebo gel

INTERVENTIONS:
Drug: nitric oxide gel — 1. st gel: sodium nitrites,BID local use X 28 days
  2. nd gel: maleic/ascorbic acids ,BID local use X 28 days
  Arms: nitric oxide gel
Drug: placebo gel — placebo gel,BID local use X 28 days
  Arms: Placebo gel

SUMMARY:
This is a randomized, double-blind, placebo-controlled, 2-period crossover, 12-week trial to be conducted in 50 subjects with painful diabetic neuropathy. The objective of this trial is to assess the safety and efficacy of NO gel, a NO donor, as compared with a placebo gel, in symptom relief of subjects with painful diabetic neuropathy.

DETAILED DESCRIPTION:
Neuropathic pain is a common symptom of diabetic neuropathy, and predominantly involves the lower limbs. Current strategies for the management of painful diabetic neuropathy include improved glycemic control, use of analgesics and addition of tricyclic antidepressants and anticonvulsants. However, many patients experience unsatisfactory responses and some undesired side effects. Considerable evidence implicates impaired nitric oxide synthesis plays an important role in the pathogenesis of diabetic neuropathic pain. Several small studies have shown that topical nitroglycerin ointment has local vasodilating properties, and a previous study has demonstrated that isosorbide dinitrate in spray form as a nitric oxide donor relieved some neuropathic symptoms in patients with painful diabetic neuropathy. Based on the findings, the investigators hypothesize that nitric oxide gel could be used as an alternative pain-relieving agent for patients with resistant diabetic neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects>=30 and<=80 years of age.
2. Subjects with type 1 or type 2 diabetes mellitus with painful diabetic neuropathy.
3. Subjects without undergoing treatment for painful diabetic neuropathy or with treatment for at least 3 months but still presenting neuropathic pain prior to randomization.
4. Subjects who are healthy without any serious diseases that require hospitalization during the study period.
5. Subjects who are capable of understanding and having signed the Informed Consent Form after detailed description of the treatment procedures and potential risks and benefits.

Exclusion Criteria:

1. Subjects with diagnosis of cancer and are still on active therapies.
2. Subjects with diagnosis of an active disease (e.g. hyper-or-hypothyroidism, advanced chronic renal failure, severe anemia, liver cirrhosis, active infectious disease etc.) and are still under regular treatment for this disease
3. Subjects with peripheral neuropathy caused by a known acute or chronic disease or injury
4. Subjects who are on other medications with pharmacological actions that may lead to excessive formation of nitric oxide (e.g. sublingual nitroglycerin, sildanafil etc.) or may accentuate drug effects due to excessive formation of nitric oxide.
5. Subjects with severe peripheral artery disease leading to absence of foot pulses.
6. Subjects with erratic glycemic control (HbA1c 12).
7. Subjects with an active foot ulceration or infection.
8. Subjects with any known allergic reaction to any ingredient in the 2 gel preparations.
9. Subjects who have been enrolled into any clinical study in the preceding 3 months prior to randomization.
10. Subjects with current substance or alcohol abuse that in the opinion of the investigator would interfere with compliance or with interpretation of the study result
11. Female subject of childbearing potential who is lactating or has positive urine pregnancy test at V0 or refuses to adop reliable method of contraception during the study.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-07; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Neuopathic Pain Scale | 12 weeks

SECONDARY OUTCOMES:
vascular duplex parameters | 12 weeks
the likelihood of reusing the nitric oxide gel recorded | 12weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Chu Chen, M.D., Principal Investigator — China Medical University Hospital; Ching-Chu Chen, M.D, Study Director — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan